CLINICAL TRIAL: NCT03687346
Title: Biological Risk Factors for Onset of Binge Eating and Compensatory Behaviors
Status: Completed | Type: Observational
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: BioRF Pilot
Record Dates: First submitted 2018-09-21; First posted 2018-09-27 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Eating Disorder
Keywords: fMRI; Eating disorder; adolescent
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High Risk Group: Parental history of eating pathology
- Low Risk Group: No parental history of eating pathology

SUMMARY:
The purpose of this proposed project is to test whether several biological factors (such as elevated brain reward region and attention region response to high-calorie foods, weaker inhibitory region response to high-calorie foods, habitual caloric deprivation, and elevated limbic region responsivity) increase the risk of problematic eating (bingeing and purging) in female adolescents.

DETAILED DESCRIPTION:
Participants will be adolescent girls aged 13-16, some of whom will have parental history of eating pathology. Participants will be recruited from the general population but their age, gender, and the presence of parental lifetime eating pathology will create a high-risk sample. The goals of the proposed project are to (1) conduct a prospective high-risk study to test whether proposed biological risk factors predict the future onset of core ED symptoms (e.g., binge eating, compensatory behaviors); (2) test hypotheses regarding how these biological risk factors and established self-report ED risk factors may work together to predict ED behavior onset; (3) examine if certain biological factors account for the effects of certain established self-reported ED risk factors (e.g., elevated brain response to thin models accounts for the effect of questionnaire-measured thin-ideal internalization). The participants will complete a baseline assessment and then follow-ups assessments over a span of three years. In addition, participants will complete one fMRI scan after the first assessment.

During the COVID-19 shelter-at-home order, the investigators will not measure in person only outcomes including fMRI scans, height and weight measurement for BMI calculation nor IAT computer paradigms for all participants that have assessments due during this order.

ELIGIBILITY:
* Inclusion Criteria:

  * Female
  * Aged 13-16 years
* Exclusion Criteria:

  * Adolescents who report functional magnetic resonance imaging (fMRI) contraindications
  * Current Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) substance abuse disorder, eating disorder (ED), conduct disorder, attention deficit hyperactivity disorder (ADHD), or bipolar disorder
  * Weekly or greater use of psychoactive drugs (e.g., analgesics, cocaine, marijuana)
  * Serious medical complications (e.g., cancer, diabetes)
  * History of head injury
  * Relevant food allergies
  * BMI > 35

Ages: 13 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change in binge eating behaviors using the EDDI | 6 months, 1 year, 2 year, and 3 year follow-up
  Eating Disorder Diagnostic Interview (EDDI)
Change in compensatory behaviors using the EDDI | 6 months, 1 year, 2 year, and 3 year follow-up
  Eating Disorder Diagnostic Interview (EDDI)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, Ph.D., Principal Investigator — Stanford University
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

REFERENCES:
- [Derived] Stice E, Yokum S, Rohde P, Cloud K, Desjardins CD. Comparing healthy adolescent females with and without parental history of eating pathology on neural responsivity to food and thin models and other potential risk factors. J Abnorm Psychol. 2021 Aug;130(6):608-619. doi: 10.1037/abn0000686. PMID 34553956